CLINICAL TRIAL: NCT02318368
Title: A Phase 2, Multicenter, Randomized, Double-blind Study of Ficlatuzumab Plus Erlotinib Versus Placebo Plus Erlotinib in Subjects Who Have Previously Untreated Metastatic, EGFR-mutated Non-small Cell Lung Cancer (NSCLC) and BDX004 Positive Label
Brief Title: A Phase 2, Study of Ficlatuzumab Plus Erlotinib vs. Placebo Plus Erlotinib in Subjects With Previously Untreated Metastatic, EGFR-mutated NSCLC and BDX004 Positive Label
Acronym: FOCAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AV-299-14-206
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ficlatuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ficlatuzumab plus erlotinib (Experimental): 150 mg Erlotinib orally once daily starting on Day 1 of Cycle 1 with 20 mg/kg Ficlatuzumab administered intravenously once every 2 weeks on Day 1 and Day 15 of each 28 day cycle.
  Interventions: Drug: Ficlatuzumab; Drug: Erlotinib
- Placebo plus erlotinib (Active Comparator): 150 mg Erlotinib orally once daily starting on Day 1 of Cycle 1 with Placebo administered intravenously once every 2 weeks on Day 1 and Day 15 of each 28 day cycle.
  Interventions: Drug: Erlotinib; Drug: placebo

INTERVENTIONS:
Drug: Ficlatuzumab
  Other Names: Ficla
  Arms: Ficlatuzumab plus erlotinib
Drug: Erlotinib
  Other Names: Erlotinib hydrochloride
Drug: placebo
  Arms: Placebo plus erlotinib

SUMMARY:
Phase 2 multicenter, controlled, randomized, double-blind study to evaluate the efficacy and safety of ficlatuzumab versus placebo when administered with erlotinib in subjects with previously untreated metastatic EGFR-mutated NSCLC and BDX004 Positive Label.

DETAILED DESCRIPTION:
This is a Phase 2 multicenter, controlled, randomized, double-blind study to evaluate the efficacy and safety of ficlatuzumab versus placebo when administered with erlotinib in subjects with previously untreated metastatic EGFR-mutated NSCLC and BDX004 Positive Label.

Prior to screening, subjects will have tested positive for a sensitizing EGFR mutation to determine eligibility for treatment with erlotinib. During screening, subject serum samples will be tested using the investigational companion diagnostic (BDX004) test. Only those subjects who have a BDX004 Positive Label will be enrolled. Subject randomization will be stratified by EGFR mutation type and smoking status (ever versus never smokers). Subjects will be designated as never smokers if they have smoked less than 100 cigarettes in their lifetime. Radiographic tumor assessment, to include CT or MRI of chest and abdomen, will be performed every 4 weeks for the first 8 cycles, and every 8 weeks thereafter, using the same imaging modality per subject. Safety assessments will be performed on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria

* Histologically and/or cytologically confirmed primary diagnosis of Stage IV NSCLC (according to American Joint Committee on Cancer [AJCC] 7th edition lung cancer staging criteria).
* Measurable disease according to RECIST v.1.1.
* An EGFR exon 19 deletion and/or an exon 21 (L858R) substitution mutation.
* BDX004 Positive Label.
* Have received no prior systemic chemotherapy, immunotherapy, targeted therapy, or biologic therapy for metastatic NSCLC. Subjects may have previously been treated with postoperative adjuvant chemotherapy for early stage lung cancer or chemo radiotherapy for locally advanced disease provided this was completed at least 6 months prior to enrollment. No prior EGFR TKI therapy is allowed for any stage of NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Exclusion Criteria
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent or erlotinib.
* History of known brain metastases.
* Prior treatment with any other investigational drug or biologic agent within 5 half lives prior to randomization, or any investigational device within 2 weeks prior to randomization.
* Any unresolved toxicity from previous radiation therapy.
* Significant cardiovascular disease, including:

  * Echocardiogram (ECHO) or multiple gated acquisition (MUGA) showing left ventricular ejection fraction of less than 55%.
  * Cardiac failure New York Heart Association class III or IV.
  * Myocardial infarction, severe or unstable angina within 6 months prior to randomization.
  * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation).
  * Significant thrombotic or embolic events within 3 months prior to randomization (significant thrombotic or embolic events include but are not limited to stroke or transient ischemic attack).
  * Any uncontrolled or severe cardiovascular disease.
* History of prior malignancy within 3 years prior to randomization (except for adequately treated non-melanoma skin cancer, carcinoma in situ of the breast or cervix, superficial bladder cancer, or early stage prostate cancer, without evidence of recurrence).
* Radiographic evidence of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Needle, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (47):
- United States (13):
  - UCSF Fresno, Fresno, California
  - Torrance Memorial Medical Center, Redondo Beach, California
  - Boca Raton Regional Hospital Lynn Cancer Institute, Boca Raton, Florida
  - University of Miami Sylvester Comprehensive Cancer Center Deerfield Beach, Deerfield Beach, Florida
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Cancer Center of Acadiana, Lafayette, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Valley Medical Group, Paramus, New Jersey
  - Queens Hospital Cancer Center, Jamaica, New York
  - Aultman Hospital, Canton, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - UPMC Cancer Center Cancer, Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (10):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Icon Cancer Care, Southport, Queensland
  - Princess Alexandra Hospital, Wolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Eastern Health, Box Hill, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Ballarat Oncology and Haematology, Wendouree, Victoria
- Hong Kong (2):
  - Tuen Mun Hospital, Tuenmen, N.T
  - Queen Mary Hospital, Pok Fu Lam
- Italy (8):
  - AO G.Rummo, Benevento
  - Policlinico S.Orsola Malpighi, Bologna
  - Istituti Ospitalieri di Cremona - Oncologia, Cremona
  - U.O.C. Oncologia, Lucca
  - IRCCS Ospedale S.Raffaele, Milan
  - Fondazione Salvatore Maugeri, Pavia
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Ospedale Treviglio-Caravaggio, Treviglio BG
- Singapore (2):
  - John Hopkins Singapore International Medical Center, Central Singapore
  - National Cancer Centre, Singapore
- South Korea (5):
  - Korea University Guro Hospital, Guro-gu, Seoul
  - Chungbuk National University Hospital, Chungcheongbuk-do
  - Chonnam National University Hwasun Hospital, Jeonnam
  - Severance Hospital, Yonsei Uni, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (7):
  - Chung Shan Medical University, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Medical University, Taipei
  - Chang Gung Medical Foundation, Taoyuan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were enrolled in 9 sites in the United States, Australia, Hong Kong, Italy, Singapore, Korea, and Taiwan. The Sponsor terminated Study AV-299-14-206, effective 14-Sep-2016, after determining that enrollment of participants was much lower than expected.
Pre-assignment Details: Prior to screening, subjects who have tested positive for a sensitizing Epidermal growth factor receptor (EGFR) mutation to determine eligibility for treatment with erlotinib. All participants underwent inclusion exclusion criteria assessment and all eligible participants signed the informed consent before undergoing any study-related procedures.
Groups:
- Ficlatuzumab Plus Erlotinib: Participants received 150 mg Erlotinib orally once daily starting on Day 1 of Cycle 1 with 20 mg/kg Ficlatuzumab administered intravenously once every 2 weeks on Day 1 and Day 15 of each 28 day cycle.
- Placebo Plus Erlotinib: Participants received 150 mg Erlotinib orally once daily starting on Day 1 of Cycle 1 with Placebo administered intravenously once every 2 weeks on Day 1 and Day 15 of each 28 day cycle.
Period: Overall Study
Arm/Group | Ficlatuzumab Plus Erlotinib | Placebo Plus Erlotinib
Started | 7 | 3
Completed | 0 | 0
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study terminated by the sponsor | 5 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ficlatuzumab Plus Erlotinib | Placebo Plus Erlotinib | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the time from the date of randomization to the date of the first objective documentation of radiographic disease progression or death due to any cause, whichever occurs first.
Time Frame: Approximately 24 months
Population: The study was terminated prior to completing enrollment; after determining that enrollment of subjects was much lower than expected, no data was collected for this outcome measure.
Arm/Group | Ficlatuzumab Plus Erlotinib | Placebo Plus Erlotinib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: To evaluate Safety and tolerability of ficlatuzumab plus erlotinib versus placebo plus erlotinib in subjects who have previously untreated metastatic EGFR-mutated NSCLC and a BDX004 Positive Label.
Time Frame: Approximately 24 months
Population: All participants who received one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Ficlatuzumab Plus Erlotinib | Placebo Plus Erlotinib
Number analyzed (Participants) | 7 | 3
Participants
  Patients with Treatment-Emergent Adverse Events | 7 | 3
  Patients with Serious Adverse Events | 3 | 1
  Patients with grade 5 TEAEs | 0 | 0
  Patients with grade 3 or 4 TEAEs | 4 | 1
  Patients permanently discontinued | 2 | 0
  Patients with dose reduction or interruption | 3 | 0

ADVERSE EVENTS:
Time Frame: Approximately 24 months
Description: An AEs is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In addition abnormal findings in vitals signs, resting 12-lead pECGs (electrocardiography), continuous dECGs, cardiac telemetry and spirometry were reported as AEs.
Arm/Group | Ficlatuzumab Plus Erlotinib | Placebo Plus Erlotinib
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ficlatuzumab Plus Erlotinib (N=7) | Placebo Plus Erlotinib (N=3)
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ficlatuzumab Plus Erlotinib (N=7) | Placebo Plus Erlotinib (N=3)
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Paronychia (Infections and infestations) | 1 | 1
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The Sponsor terminated Study AV-299-14-206 before enrollment was completed, effective 14-Sep- 2016, after determining that enrollment of subjects was much lower than expected, and that timely completion of the study was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No